CLINICAL TRIAL: NCT02455622
Title: A Long-Term, Open-Label, Multicenter, Phase IV Study to Assess Longitudinal Changes on Height and Weight in Patients With MPS II Who Are Receiving Elaprase and Started Treatment With Elaprase at <6 Years of Age
Brief Title: Long-term Evaluation on Height and Weight in Patients With MPS II Who Started Treatment at < 6 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP-ELA-401; 2014-004804-31 (EudraCT Number)
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II | interventions — idursulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enrolled Patients (Experimental): Patients who are receiving treatment with Elaprase in this study (SHP-ELA-401), who are <6 years of age, and were previously treatment-naïve. Patients who are not enrolled in this study (SHP-ELA-401) but are enrolled in the Hunter Outcome Survey (HOS) patient registry and were < 6 years of age at start of Elaprase treatment. While not enrolled in the present Study SHP-ELA-401, their height and weight data from HOS will be utilized in the Primary Growth Analysis for this study.
  Interventions: Drug: Elaprase for intravenous (IV) infusion

INTERVENTIONS:
Drug: Elaprase for intravenous (IV) infusion — Patients enrolled in this study will receive once-weekly IV infusions of Elaprase at a dose of 0.5 mg/kg and will be followed for a minimum of 5 years after initiation of Elaprase treatment, or until they reach their 10th birthday, whichever is longer.Height and weight data from HOS will be utilized in the Primary Growth Analysis for this study.
  Other Names: Idursulfase

SUMMARY:
This long-term study will provide Elaprase treatment to children enrolled in this study and will utilize data from both enrolled patients and Hunter Outcome Survey (HOS) patient registry data to conduct the primary growth analysis to assess changes in height and weight in patients with Mucopolysaccharidosis II (Hunter syndrome) MPS II.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Prospective Patient Group

  1. The patient is male.
  2. The patient is Elaprase-naïve at study entry.
  3. The patient must have a documented diagnosis of MPS II. Of the 3 criteria below, the combinations (3a AND 3b) or (3a AND 3c) will be accepted as diagnostic of MPS II:

     1. The patient has a deficiency in I2S enzyme activity of ≤10% of the lower limit of the normal range as measured in plasma, fibroblasts, or leukocytes (based on the reference laboratory's normal range). AND
     2. The patient has a documented mutation in the I2S gene. OR
     3. The patient has a normal enzyme activity level of one other sulfatase as measured in plasma, fibroblasts, or leukocytes (based on the normal range of measuring laboratory).
  4. The patient will be <6 years of age at the start of Elaprase treatment.
  5. The patient, patient's parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form after all relevant aspects of the study have been explained and discussed. Consent of the patient's parent(s) or legally authorized guardian(s) and the patient's assent, as relevant, must be obtained.

Group 2: Retrospective Data Inclusion Criteria:

Retrospective Patient Group patients will be enrolled in HOS and not Study SHP-ELA-401; however, their growth data may be included in the analysis for Study SHP-ELA-401 if the following data inclusion criteria are met.

1. The patient is male.
2. The patient is enrolled in HOS.
3. The patient was <6 years of age at the start of Elaprase treatment.
4. The patient received Elaprase weekly treatment for at least 5 years.
5. The patient had a height assessment and a weight assessment documented within 3 months before or after Elaprase treatment start.
6. The patient has had annual height and weight assessments from start of Elaprase through age 10 years.
7. The patient, patient's parent(s), or legally authorized guardian(s) agree(s) to data collection.
8. The patient, patient's parent(s), or legally authorized guardian(s) must have signed an IRB/IEC-approved informed consent form after all relevant aspects of the HOS study have been explained and discussed. Consent of the patient's parent(s) or legally authorized guardian(s) and the patient's assent, as relevant, must be obtained.

Exclusion Criteria:

* Group 1: Prospective Patient Group

  1. The patient has received treatment with any investigational drug or device within the 30 days prior to study entry.
  2. The patient has received or is receiving treatment with idursulfase-IT.
  3. The patient has received growth hormones, a cord blood infusion, or a bone marrow transplant at any time.
  4. The patient has received blood product transfusions within 90 days prior to Screening.
  5. The patient is unable to comply with the protocol as determined by the Investigator.

Group 2: Retrospective Data Exclusion Criteria:

HOS patients that meet the following criteria are not eligible to be included into the Study SHP-ELA-401 Primary Growth Analysis:

1. Patient was treated with growth hormone or other medications or interventions intended to promote growth in the time period covered by the analysis.

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Change in height | Screening to End-of-Study (5-10 years)
Change in weight Z-scores | Screening to End-of-Study (5-10 years)
Change in neurological examination to evaluate long-term safety in patient | Screening to End-of-Study (5-10 years)
Number of participants with adverse events as measured by type, severity, and relationship to treatment | Screening to End-of-Study (5-10 years)
Change in clinical laboratory testings as measured by urinalysis to evaluate long-term safety in patients | Screening to End-of-Study (5-10 years)
Change in clinical laboratory testings as measured by serum chemistry to evaluate long-term safety in patients | Screening to End-of-Study (5-10 years)
Change in clinical laboratory testings as measured by hematology to evaluate long-term safety in patients | Screening to End-of-Study (5-10 years)

SECONDARY OUTCOMES:
Urinary glycosaminoglycans (uGAG) levels normalized to urine creatinine | Screening to End-of-Study (5-10 years)
Normalized uGAG divided by upper limit of normal for age (uGAG/ULN) every 12 months | Baseline to End-of-Study (5-10 years)
Joint mobility, as measured by Joint Range of Motion (JROM) scores, including global, upper-limb, and lower-limb joint scores | Screening to End-of-Study (5-10 years)
Distance walked, as measured by the Six Minute Walk Test (6MWT) | Screening to End-of-Study (5-10 years)
Quality of Life, as measured by the Hunter-Syndrome Functional Outcome in Clinical Understanding Scale | Screening to End-of-Study (5-10 years)
Impact of illness on ability to function in daily life, as measured by the Childhood Health Assessment Questionnaire (CHAQ Parent Report) | Screening to End-of-Study (5-10 years)
Adaptive behavior, as measured by the Vineland Adaptive Behavior Scales (VABS II) | Screening to End-of-Study (5-10 years)
Change in anti-idursulfase antibodies in serum | Screening to End-of-Study (5-10 years)
  number and percentage of patients testing anti-idursulfase antibody positive and negative at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (8):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States
- Hospital Infantil Dr Robert Reid Cabral, Santo Domingo, Dominican Republic
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Germany
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia
- Philippine General Hospital, Manila, Philippines
- Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade, Serbia
- Chulalongkorn University, Bangkok, Thailand
- National Pediatrics Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f6b5fe94db2bf003ab47b2e